CLINICAL TRIAL: NCT03040609
Title: Development of a Visio-behavioral Scale to Evaluate Visual Abilities of Patients With Profound Multiple Intellectual Disabilities (PLH-Vision)
Acronym: PLH-Vision
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P140712; RCB: 2016-A00278-43 (Other: ANSM)
Record Dates: First submitted 2016-12-12; First posted 2017-02-02 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-02

CONDITIONS: Profound Multiple Intellectual Disabilities
Keywords: Profound Multiple Intellectual Disabilities; Visual-Behavioral Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: The duration of follow-up of group 1 in the study is 1 day.
  Interventions: Behavioral: Visual-behavioral Scale at day 1; Behavioral: Test-retest at the end of 2 weeks; Behavioral: Test at 6 months
- Group 2: The duration of follow-up of group 2 in the study is 2 weeks.
  Interventions: Behavioral: Test-retest at the end of 2 weeks; Behavioral: Test at 6 months
- Group 3: The duration of follow-up of group 3 in the study is 6 months.
  Interventions: Behavioral: Test at 6 months

INTERVENTIONS:
Behavioral: Visual-behavioral Scale at day 1 — To perform the classification with the scale by caregiver.
  Groups: Group 1
Behavioral: Test-retest at the end of 2 weeks — To perform the classification with the scale by orthoptist at the end of 2 weeks
  Groups: Group 1; Group 2
Behavioral: Test at 6 months — To perform the classification with the scale by orthoptist at the end 6 months.

SUMMARY:
The main objective of this study is to develop and validate a visio-behavioral scale of visual abilities for subjects with profound multiple intellectual disabilities.

The secondary objectives of the study are:

* to validate the structure of the scale.
* to evaluate the reproducibility of scale with the intra- and inter-examiners, and the influence of the different professions of examiners.
* to evaluate the feasibility of visio-behavioral scale.
* to evaluate the sensitivity to change.
* to study the uniformity of use of the scale depending on the type of patients (age, disability level, pathology).
* to study the prevalence of the visual disorder in profound multiple intellectual disabilities subjects.

DETAILED DESCRIPTION:
This study includes 3 phases:

* Elaboration of a list of behavioral items by a group of multi-disciplinary expertise (physicians, nurses, caregivers, ophthalmologies, orthoptists) based on their clinical experiences.
* Development of the scale based on the sample obtained by a prospective multicenter research trial.
* Validation of the sample obtained by a prospective transversal multicenter study.

This study will be performed in 5 centers in France. The enrollment of patients planned for 24 months targeting 310 patients. The duration of follow-up of the study for each patient will be varied according to the group of patients, il will be 1 day for group 1, 2 weeks for group 2, or 6 months for group 3.

ELIGIBILITY:
Inclusion Criteria:

* Causal brain injury occurred before the age of 3 years.
* Severe or deep mental retardation as defined by DSM IV.
* Motor impairment: para / tetraparesis, hemiparesis, ataxia, or extrapyramidal motor disorders.
* Score of Gross Motor Function Classification System [Palisano 1997] is III, IV or V.
* Score of Functional Independence Measure < 55.
* Subject aged ≥3 years (because the visio-behavioral scale is not adapted for children younger than 3 years).
* Beneficiary of a social protection.
* Written consent signed by guardian or legal representative, or parents in case of a minor subject.

Exclusion Criteria:

* Acute intercurrent pathology precluding examinations.
* Patient with hypersensitivity to tropicamide, atropine or benzalkonium chloride.
* Angle closure glaucoma suspect patient.
* Patient with severe hypertension.
* Short life expectancy.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Profound multiple intellectual disabilities patients aged 3 years or older.
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Concordance of classification | throughout the study: 31 months
  Statistical analysis: concordance between the classification obtained by caregiver with the scale, and the classification obtained by orthoptist-ophthalmology.

SECONDARY OUTCOMES:
Structure of the scale | throughout the study: 31 months
  Statistical analysis to validate the structure of the scale.
Reproducibility of scale | throughout the study: 31 months
  Statistical analysis to evaluate the reproducibility of scale with the intra- and inter-examiners, and the influence of the different professions of examiners.
Feasibility of visio-behavioral scale | throughout the study: 31 months
  Statistical analysis to evaluate by the proportion of patients who have the complet examination, the average of time to all examens, the tolerance data.
  feasibility of visio-behavioral scale.
Sensitivity to change | throughout the study: 31 months
  Statistical analysis to evaluate the sensitivity to change.
Uniformity of use of the scale | throughout the study: 31 months
  Statistical analysis to assess the uniformity of use of the scale depending on the type of patients (age, disability level, pathology).
Prevalence of the visual disorder | throughout the study: 31 months
  Statistical analysis to study the prevalence of the visual disorder in profound multiple intellectual disabilities subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine ROUSSEAU, MD, Principal Investigator — AP-HP, Hôpital San Salvadour, 83407 Hyères; Soizic CHARBONNIER, Orthoptist, Study Chair — Cabinet du Lycée
Locations (1):
- Hôpital San Salvadour, Hyères, Var, France

IPD SHARING:
Plan to Share IPD: No